CLINICAL TRIAL: NCT02890602
Title: A Phase Ⅱ Study of Erythropoietin for Management of Anemia Caused by Chemotherapy in Patients With Diffuse Large B-cell Lymphoma
Brief Title: Erythropoietin for Management of Anemia Caused by Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kosin University Gospel Hospital (Other)
Responsible Party: Principal Investigator, Ho Sup Lee, MD, PhD. associate professor, Division of hematology-Oncology, Kosin University Gospel Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EPOMA
Record Dates: First submitted 2016-08-18; First posted 2016-09-07 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Darbepoetin alfa; R-CHOP protocol; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Darbepoietin alfa (Experimental): Hemoglobin level will be checked at every cycle's day 0 or 1(1cycle is 21days) after starting Darbepoietin alfa. It will be applied to chemotherapy until increment of hemoglobin 12.0 g/dL.
  Interventions: Drug: Darbepoetin alfa; Drug: R-CHOP

INTERVENTIONS:
Drug: Darbepoetin alfa — Darbepoietin alfa will be administered subcutaneously at a fixed dose of 360㎍. If it is impossible, administration by intravenous infusion is okay.
  Other Names: Nesp
Drug: R-CHOP — R-CHOP regimen is a practical procedure in patients with Diffuse Large B-cell Lymphoma. Darbepoietin alfa will be administered to these patients.
  Other Names: Rituximab, Cyclophosphamide, Adriamycin, Vincristine, Prednisolone

SUMMARY:
This is a phase Ⅱ study of erythropoietin for management of anemia caused by chemotherapy in patients with Diffuse Large B-cell Lymphoma. The investigators want to investigate hematopoietic response of darbepoietin alfa and the quality of life assessment of increasement of hemoglobin.

DETAILED DESCRIPTION:
Darbepoietin alfa may cause the body to make more red blood cells. They are used to treat anemia caused by chemotherapy in patients with malignant lymphoma. Darbepoietin will be applied to R-CHOP(Rituximab, Cyclophosphamide, Adriamycin, Vincristine, Prednisolone) chemotherapy every 21days ± 2days with fixed 360㎍. It will be applied to chemotherapy until increment of hemoglobin 12.0g/dL. If the hemoglobin level exceeds 12.0g/dL, administration of darbepoietin will be temporarily stopped.

And, the questionnaire of the quality of life will be conducted at the baseline, after 2th darbepoietin alfa administration, at study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diffuse large B cell lymphoma treated with R-CHOP(Rituximab, Cyclophosphamide, Adriamycin, Vincristine, Prednisolone) chemotherapy
2. hemoglobin < 10.0 g/dL are shown at least 3 cycles after starting R-CHOP(Rituximab, Cyclophosphamide, Adriamycin, Vincristine, Prednisolone)
3. Currently receiving or planning to receive at least 4 times of darbepoetin
4. Age > 18 years
5. ECOG(Eastern Cooperative Oncology Group) performance status 0-2
6. Bilirubin < 2 times upper limit of normal
7. ALT(alanine aminotransferase) or AST(aspartate aminotransferase) < 5 times upper limit of normal
8. Creatinine < 2 times upper limit of normal
9. HIV negative
10. Ferritin > 20 mcg/L (i.e., not obviously iron deficient)
11. Can read Quality of life as measured by Functional Assessment of Cancer Therapy Scales for Anemia
12. Agree with informed consent

Exclusion Criteria:

1. Received radiation therapy at least 4 weeks before starting chemotherapy
2. serious pre-existing medical condition (e.g., cardiac failure [New York Heart Association Class III or IV, or left ventricular ejection fraction <50%], active peptic ulceration, uncontrolled diabetes mellitus, or acute diffuse infiltrative pulmonary disease)
3. uncontrolled hypertension, defined as systolic blood pressure (BP) ≥ 180 mm Hg and/or diastolic BP ≥ 100 mm Hg, despite medical therapy
4. arrhythmia NCI CTCAE grade ≥ 2
5. History of previously treated seizures allowed provided the patient has been seizure-free for a minimum of 3 months
6. active systemic infection requiring treatment, a known diagnosis of human HIV, or active hepatitis B (hepatitis B carriers were permitted)Malignancy was treated surgically or with local radiation therapy with curative intent and the patient has been disease free for > 3 years
7. known hypersensitivity to darbepoetin alfa
8. pregnant or nursing and Negative pregnancy test
9. previous diagnosis of another malignancy with radiographic or biochemical evidence of residual disease (except completely resected basal cell carcinoma, squamous cell carcinoma of the skin, or an in-situ malignancy)
10. combined iron deficiency anemia
11. received erythropoietin at least one months before starting darbepoetin
12. considered autologous stem cell transplantation before finish 6 cycles of chemotherapy
13. untreated primary or metastatic CNS(central nervous system) malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-09-01; Primary Completion 2017-11-28 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Hematopoietic response | hemoglobin level of day 21 after Darbepoietin alfa administration
  Hemoglobin level after Darbepoietin alfa administration

SECONDARY OUTCOMES:
Quality of life as measured by Functional Assessment of Cancer Therapy Scales for anemia | at baseline, Day 21 after 2th darbepoietin alfa administration, Day 21 after last darbepoietin alfa administration
Adverse events as measured by CTCAE v3.0 | From the date of first drug administration to the date of the 30th days of last drug administration.
Proportion of patients requiring red blood cell transfusions | From the date of first darbepoietin alfa administration to day 21 after last darbepoietin alfa administration
Mean time to response of hemoglobin | From the date of first darbepoietin alfa administration to day 21 after last darbepoietin alfa administration